CLINICAL TRIAL: NCT02721043
Title: Study Of Pgv001 A Multi-Peptide Therapeutic Vaccine Platform For Use In The Treatment Of Malignancies In The Adjuvant Setting
Brief Title: Safety and Immunogenicity of Personalized Genomic Vaccine to Treat Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nina Bhardwaj (Other)
Responsible Party: Sponsor-Investigator, Nina Bhardwaj, Director of Immunotherapy Program, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 15-1811
Record Dates: First submitted 2016-02-16; First posted 2016-03-28 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2020-01

CONDITIONS: Solid Tumors
Keywords: Personalized vaccine; Poly-ICLC; Immunotherapy; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Peptides; poly ICLC; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Personalized Genome Vaccine 001 (Experimental): PGV-001 (peptides + Poly-ICLC)
  Peptides: 100mcg per peptide per dose.
  Poly-ICLC (Hiltonol®, Oncovir): 1.4mg (0.7mL, 2mg/mL)
  Interventions: Biological: Peptides; Drug: Poly-ICLC; Drug: Lenalidomide

INTERVENTIONS:
Biological: Peptides — Each subject will receive ten (10) total doses of PGV001. PGV001 will be administered on study visit: v4, v6, v8, v10, v12, v14, v16, v18, v20 and v22.
  Other Names: Personalized Genome Vaccine 001; PGV 001; personalized peptide vaccine
Drug: Poly-ICLC — Each subject will receive ten additional (10) total doses of the Poly-ICLC. The additional Poly-ICLC dose will be administered on study visit: v5, v7, v9, v11, v13, v15, v17, v19, v21 and v23.
  Other Names: Hiltonol®
Drug: Lenalidomide — 10mg once daily oral dose for maintenance therapy in multiple myeloma patients.

SUMMARY:
The purpose of this study is to test the safety, tolerability, and immunogenicity of Personalized Genomic Vaccine 001 (PGV001) in subjects with advanced non-hematologic malignancies. PGV001 is a peptide vaccine that is based on a patient's own tumor sequence. Each patient's tumor is sequenced and peptides that correspond to the tumors are made. These peptides combined with the adjuvant Poly-ICLC (Hiltonol®, Oncovir) make PGV001. The adjuvant Poly-ICLC is added to boost the immune response to the peptides and together will expand immune cells to target cancer.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have a histologically or cytological-proven diagnosis of one of the following malignancies:

  1. Oral, oropharyngeal, hypopharyngeal or laryngeal squamous cell carcinoma
  2. Non-small cell carcinoma of the bronchus and/or lung
  3. Ductal or lobular carcinoma of the breast
  4. Serous carcinoma of the ovary, fallopian tube, or other uterine adnexa
  5. Urothelial cell carcinoma of renal pelvis, ureter, or bladder
  6. Cutaneous squamous cell carcinoma
  7. All epithelial carcinoma of the ovary, fallopian tube, or other uterine adnexa
* The subject must be medically capable of providing the necessary tissue sample for sequencing, either by surgical resection or open-surgical or core biopsy sampling of the primary tumor.

  a. This requirement may be satisfied by providing an archival tissue sample in the form of a formalin-fixed paraffin-embedded or frozen tissue block from an earlier resection.
* The subject must have no measurable disease at the time of investigational product administration.

  1. The subject must complete all prior surgery requiring general anesthesia at least four (4) weeks before administration of the investigational product. The subject must complete all surgery requiring local/epidural anesthesia at least seventy-two (72) hours prior to administration of the investigational product.
  2. The subject must complete all prior systemic chemotherapy therapy, and all adverse events have either returned to baseline or have stabilized at least four (4) weeks prior to administration of the investigational product.
  3. The subject must complete all prior systemic radiation therapy at least four (4) weeks prior to administration of the investigational product. The subject must complete all prior focal radiation therapy at least two (2) weeks prior to the administration of the investigational agent. The subject must not have received a radiopharmaceutical within eight (8) weeks prior to the administration of the investigational product.
  4. The subject may continue hormonal therapy (i.e tamoxifen, anastrozole) during the study.
* The risk of disease recurrence with a five (5) year time period, as estimated by the treating physician, must be greater than or equal thirty percent (30%).
* The subject must have a life expectancy greater than twelve (12) months at the time of screening.
* The subject must have a performance status of 0-1 as determined by criteria set forward by the Eastern Cooperative Oncology Group.
* The subject must have at the time of screening acceptable hematologic, hepatic, and renal function, defined by the following:

  1. Absolute neutrophil count ≥ 1000/mm3
  2. Platelet count ≥ 50,000/mm3,
  3. Creatinine ≤ 2.5 mg/dL,
  4. Total bilirubin ≤ 1.5 mg/dL,
  5. Transaminases ≤ 2 times above the upper limits of the institutional normal.
  6. INR<2 if off of anticoagulation. Patients on anticoagulation therapy with an INR>2 may be enrolled at the discretion of the investigator if they have not had any episodes of severe hemorrhage.
* The subject must be 18 years of age or older.
* The subject must be deemed competent to give informed consent.
* The subject must agree to use two effective forms of contraception beginning at least four (4) weeks prior to study entry, and continuing to do so for the duration of their participation in the study.

Exclusion Criteria:

* The subject has metastatic disease at the time of screening.
* The subject has a history of unrelated neoplastic disease, which has been deemed active within thirty-six (36) months of the screening evaluation, with the exception of the following:

  1. Non-invasive non-melanoma skin cancer such as superficial basal cell carcinoma or squamous cell carcinoma.
  2. In female subjects: High-grade or low-grade squamous intraepithelial lesions or equivalent cervical lesions
  3. In male subjects: tumors of the prostate with a combined Gleason Score ≤ 7
* The subject has a prior history of unrelated neoplastic disease, and has received systemic therapy for the secondary malignancy within the twelve (12) month period preceding the screening evaluation.
* The subject has a history of Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome (HIV/AIDS), Chronic hepatitis B or hepatitis C or is otherwise reasonably suspected to meet criteria for the diagnosis of a known congenital or acquired disorder causing systemic immunosuppression.
* The subject has a history of, or is reasonably suspected to meet criteria for the diagnosis of a known congenital or acquired disorder causing systemic immunosuppression; or the subject is currently receiving any drug or supplement which is known to be associated with systemic immune suppression including those drugs which are prescribed for solid organ or stem cell transplant, autoimmune/inflammatory disorders, or other related medical conditions.
* The subject has a history of, or is reasonably suspected to meet criteria for the diagnosis of a systemic auto-immune/inflammatory disease or other autoimmune disorder with the exception of:

  a. Vitiligo
* The subject has a history of anaphylaxis or other serious adverse reactions relating to administration of any components of the investigational product.
* The subject has a history of serious allergic reaction to any substance, resulting in hospitalization or requiring other emergent medical attention.
* The subject has a history of advanced cardiac, hepatic or renal disease or other chronic illness.
* The subject has been diagnosed and treated at an external facility, and the resulting tissue specimen is of insufficient quality such that it precludes clinical sequencing or any other necessary study procedure, and the subject is unwilling to undergo an additional biopsy procedure.
* The subject is less than eighteen (18) years of age, or otherwise unable to give informed consent due to minor status.
* The subject is a prisoner, as defined by [45 CFR 46.303(c)].
* The subject is cognitively impaired, and unable to give informed consent.
* The subject is pregnant, as defined by a presumptive sign of pregnancy such as missed menses or a positive pregnancy test [45 CFR 46.203(b)].

Note: The effects of the investigational product on the developing human fetus are unknown. Female subjects of childbearing potential are required to have a negative qualitative serum pregnancy test at the time of enrollment and within twenty-four (24) hours prior to the first dose of the investigational product.

1. Female subject of childbearing potential is defined as follows:

   1. Subject with regular menses
   2. Subject with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
   3. Subject with history of tubal ligation
2. Female subject not of childbearing potential is defined as follows:

   1. Subject who has undergone hysterectomy and/or bilateral oophorectomy.
   2. Subject who is post-menopausal, which is defined as amenorrhea for at least one (1) year in a female subject who is greater than forty-five (>45) years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-04; Primary Completion 2019-11-12 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | up to day 42
  toxicity will be measured by severity of Adverse events with toxicity grading defined by Cancer Therapy Evaluation Program's (CTEP) v4.0 of National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) scale
Toxicity grading using CTCAE scale | one year
  safety will be measured by number of Adverse events with toxicity grading defined by Cancer Therapy Evaluation Program's (CTEP) v4.0 of National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) scale

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No